CLINICAL TRIAL: NCT00560404
Title: A Randomized, Open Label Study to Compare the Effect of Once Monthly Administration of Subcutaneous Mircera Versus Epoetin Alfa on Maintenance of Hemoglobin Levels, Safety and Tolerability in Dialysis Patients With Chronic Renal Anemia.
Brief Title: A Study of Subcutaneous Mircera for the Maintenance Treatment of Dialysis Patients With Chronic Renal Anemia.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ML21208
Record Dates: First submitted 2007-11-16; First posted 2007-11-19 (Estimated); Results first posted 2016-04-12 (Estimated); Last update posted 2025-09-11 (Actual); Status verified 2025-08

CONDITIONS: Anemia
MeSH Terms: conditions — Anemia | interventions — continuous erythropoietin receptor activator; Epoetin Alfa

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: methoxy polyethylene glycol-epoetin beta [Mircera]
- 2 (Active Comparator)
  Interventions: Drug: Epoetin alfa

INTERVENTIONS:
Drug: methoxy polyethylene glycol-epoetin beta [Mircera] — 120, 200 or 360 micrograms sc monthly (starting dose)
  Arms: 1
Drug: Epoetin alfa — As prescribed
  Arms: 2

SUMMARY:
This 2 arm study will compare the efficacy and safety of monthly administration of subcutaneous Mircera versus epoetin alfa for the maintenance of hemoglobin levels in dialysis patients with chronic renal anemia. Patients currently receiving maintenance treatment with epoetin alfa will be randomized to receive either monthly injections of Mircera with a starting dose (120, 200 or 360 micrograms) derived from the dose of epoetin alfa they were receiving in the week preceding study start, or to continue on epoetin alfa treatment. The anticipated time on study treatment is 3-12 months, and the target sample size is 100-500 individuals.

ELIGIBILITY:
Inclusion Criteria:

* adult patients, >=18 years of age;
* chronic renal anemia;
* regular hemodialysis with the same schedule of dialysis for >=12 weeks;
* maintenance therapy with subcutaneous epoetin alfa at the same administration interval for 4 weeks.

Exclusion Criteria:

* transfusion of red blood cells during previous 2 months;
* poorly controlled hypertension requiring interruption of epoetin alfa in previous 6 months;
* acute or chronic bleeding;
* active malignant disease (except non-melanoma skin cancer).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 233 (Actual)
Dates: Start 2008-04; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (20):
- Brazil (20):
  - Belo Horizonte
  - Brasília
  - Campinas
  - Campo Grande
  - Cariacica
  - Curitiba
  - Fortaleza
  - Jaboatão dos Guararapes
  - Joinville
  - Juiz de Fora
  - Londrina
  - Natal
  - Porto Alegre
  - Ribeirão Preto
  - Rio de Janeiro
  - Salvador
  - São José do Rio Preto
  - São Luís
  - São Paulo
  - Sorocaba

REFERENCES:
- [Derived] Locatelli F, Choukroun G, Truman M, Wiggenhauser A, Fliser D. Once-Monthly Continuous Erythropoietin Receptor Activator (C.E.R.A.) in Patients with Hemodialysis-Dependent Chronic Kidney Disease: Pooled Data from Phase III Trials. Adv Ther. 2016 Apr;33(4):610-25. doi: 10.1007/s12325-016-0309-6. Epub 2016 Mar 10. PMID 26965694

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 457 participants were enrolled across 24 centers in Brazil from period April 02, 2008 to July 02, 2009.
Pre-assignment Details: All participants received epoetin alpha during a four-week safety verification period. Of 457 participants, 233 eligible participants entered the treatment period.
Groups:
- C.E.R.A.: Participants received RO0503821 (Continuous Erythropoietin Receptor Activator [C.E.R.A.]) with drug dosage of 120, 200 or 360 microgram subcutaneously, every four weeks, for 36 weeks.
- Epoetin Alpha: Participants received the same total dose of epoetin alpha administrated in the last week of screening period in the study, subcutaneously, three times a week, for 36 weeks.
Period: Overall Study
Arm/Group | C.E.R.A. | Epoetin Alpha
Started | 112 | 121
Completed | 76 | 100
Not Completed | 36 | 21
Not completed — Adverse Event | 2 | 3
Not completed — Death | 3 | 3
Not completed — Protocol Violation | 12 | 7
Not completed — Administrative Reasons | 1 | 1
Not completed — Withdrew Consent | 4 | 0
Not completed — Failure to return | 1 | 2
Not completed — Other withdrawal reason | 13 | 5

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population included participants who have received at least one dose of C.E.R.A. (Week 0) and for whom data for at least one follow-up is available.
Groups:
- C.E.R.A.: Participants received C.E.R.A. with drug dosage of 120, 200 or 360 microgram subcutaneously, every four weeks, for 36 weeks.
- Total: Total of all reporting groups
Arm/Group | C.E.R.A. | Epoetin Alpha | Total
Number analyzed (Participants) | 112 | 121 | 233
Age, Continuous [Median (Full Range); unit: years] | 54.5 [22 to 81] | 53.0 [19 to 84] | 54.0 [19 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43 | 53 | 96
  Male | 69 | 68 | 137

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Maintaining Their Mean Hemoglobin Concentration Within Plus or Minus 1 Gram/Deciliter of Their Reference Hemoglobin and Between the Target Range During Efficacy Evaluation Period
Description: The target hemoglobin (Hb) range was defined as Hb concentration (gram/deciliter [g/dL]) between 10.5 and 12.5 g/dL during the efficacy evaluation period (EEP). EEP was from Week 29 to Week 36.
Time Frame: EEP (Week 29 to Week 36)
Population: Per-protocol population included participants who received at least one dose of C.E.R.A. and had data of at least one follow-up variable excluding those participants who had not adhere the inclusion/exclusion criteria, had less than 3 recorded Hb values, and received any other epoetin alpha and blood transfusion in Weeks 0 to 44.
Measure: Number; unit: percentage of participants
Arm/Group | C.E.R.A. | Epoetin Alpha
Number analyzed (Participants) | 76 | 100
percentage of participants | 50.7 | 53.0
Statistical Analysis 1: Comparison: C.E.R.A. vs Epoetin Alpha; Test type: Non-Inferiority or Equivalence — Mean Hb within target range during efficacy evaluation period within plus or minus 1 g/dL of their reference Hb and between the target range with a non-inferiority limit of -0.15; Difference of response rates = -0.02, 95% CI 2-sided [-0.25 to 0.20]

2. Secondary Outcome: Mean Change From Baseline in Hemoglobin Concentration Between Baseline and at the Efficacy Evaluation Period
Description: The Baseline (Safety Verification Period) was from Week - 4 to Week -1.
Time Frame: Baseline (Weeks -4 to 0) and at EEP (Weeks 29 to 36)
Population: The analysis was performed on ITT population.
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | C.E.R.A. | Epoetin Alpha
Number analyzed (Participants) | 112 | 121
g/dL | -0.02 (1.40) | 0.05 (1.22)

3. Secondary Outcome: Percentage of Participants Maintaining Individual Hemoglobin Concentration Within the Range of 10.5 - 12.5 Gram/Decilitre Throughout the Efficacy Evaluation Period
Description: Percentage of participants maintaining individual Hb concentration within the Hb range 10.5 - 12.5 g/dL were reported during EEP. The EEP was from Week 29 to Week 36 of the study period.
Time Frame: EEP (Weeks 29 to 36)
Population: The analysis was performed on ITT population.
Measure: Number; unit: percentage of participants
Arm/Group | C.E.R.A. | Epoetin Alpha
Number analyzed (Participants) | 112 | 121
percentage of participants | 30.9 | 39.4

4. Secondary Outcome: Mean Time Spent in Hemoglobin Range of 10.5 - 12.5 Gram/Decilitre During the Efficacy Evaluation Period
Description: Mean time to maintain Hb in the range of 10.5-12.5 g/dL during EEP is presented.
Time Frame: EEP (Week 29 to Week 36)
Population: The analysis was performed on ITT population.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | C.E.R.A. | Epoetin Alpha
Number analyzed (Participants) | 112 | 121
days | 30.4 (19.5) | 33.9 (17.0)

5. Secondary Outcome: Number of Participants Who Required Dose Adjustments During the Dose Titration Period
Description: The number of participants who required dose adjustments of C.E.R.A and epoetin alpha were reported during the Dose Titration Period (DTP). The DTP was from Week 0 to Week 28.
Time Frame: DTP (Weeks 0 to 28)
Population: The analysis was performed on ITT population.
Measure: Number; unit: participants
Arm/Group | C.E.R.A. | Epoetin Alpha
Number analyzed (Participants) | 112 | 121
participants | 88 | 98

6. Secondary Outcome: Number of Participants Who Required Dose Adjustments During the Efficacy Evaluation Period
Description: The number of participants who required dose adjustments of C.E.R.A and epoetin alpha were reported during the Efficacy Evaluation Period (EEP). The EEP was from Week 29 to Week 36.
Time Frame: EEP (Weeks 29 to 36)
Population: The analysis was performed on ITT population.
Measure: Number; unit: participants
Arm/Group | C.E.R.A. | Epoetin Alpha
Number analyzed (Participants) | 112 | 121
participants | 35 | 39

7. Secondary Outcome: Number of Participants Received Red Blood Cells Transfusions
Description: The number of participants who received at least 1 red blood cell (RBC) transfusion (packed RBC or whole blood) during the study was reported. For this study, blood transfusion was reported during the titration period. No transfusion occurred in the EEP.
Time Frame: Up to Week 28
Population: The safety analysis population included those participants who have been treated with at least one dose of the trial medication and a safety follow-up, whether withdrawn prematurely or not
Measure: Number; unit: participants
Arm/Group | C.E.R.A. | Epoetin Alpha
Number analyzed (Participants) | 112 | 121
participants | 8 | 3

8. Secondary Outcome: Mean Values of Hemoglobin Concentration at Baseline and Week 36
Description: The mean Hb concentration for each participant throughout the study was estimated. Summary data of mean values of Hb concentration at Baseline and Week 36 are presented.
Time Frame: Baseline and Week 36
Population: The analysis was performed on safety population. The "n" represents the number of participants analyzed at a specified time point.
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | C.E.R.A. | Epoetin Alpha
Number analyzed (Participants) | 112 | 121
g/dL
  Baseline, n = 112, 121 | 11.6 (0.54) | 11.6 (0.57)
  Week 36; n = 75, 98: number analyzed (Participants) | 75 | 98
  Week 36; n = 75, 98 | 11.5 (1.33) | 11.7 (1.20)

9. Secondary Outcome: Mean Values of Hematocrit at Baseline and Week 36
Description: Hematocrit is the volume percentage of red blood cells in blood. The mean hematocrit for each participant was estimated throughout the study. Summary data of mean values of Hb at Baseline and Week 36 are presented.
Time Frame: Baseline and Week 36
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: fraction
Arm/Group | C.E.R.A. | Epoetin Alpha
Number analyzed (Participants) | 112 | 121
fraction
  Hematocrit, Baseline, n = 112, 121 | 0.35 (0.02) | 0.35 (0.02)
  Hematocrit, Week 36, n = 75, 98: number analyzed (Participants) | 75 | 98
  Hematocrit, Week 36, n = 75, 98 | 0.35 (0.04) | 0.36 (0.04)

10. Secondary Outcome: Mean Values of Mean Corpuscular Volume at Baseline and Week 36
Description: Mean corpuscular volume (MCV) is the average volume of red cells. The mean MCV concentration for each participant throughout the study was estimated. Summary data of mean values of MCV concentration at Baseline and Week 36 are presented.
Time Frame: Baseline and Week 36
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: femtoliters
Arm/Group | C.E.R.A. | Epoetin Alpha
Number analyzed (Participants) | 112 | 121
femtoliters
  Baseline; n = 112, 121 | 91.9 (5.95) | 92.2 (5.26)
  Week 36; n = 74, 97: number analyzed (Participants) | 74 | 97
  Week 36; n = 74, 97 | 90.6 (6.79) | 91.6 (5.84)

11. Secondary Outcome: Mean Values of Leukocytes and Platelets Count at Baseline and Week 36
Description: The mean values of laboratory parameters: leukocytes and platelets count for each participant was estimated throughout the study. Summary data of mean values of leukocytes and platelets count at Baseline and Week 36 are presented.
Time Frame: Baseline and Week 36
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: 10^9/Litre
Arm/Group | C.E.R.A. | Epoetin Alpha
Number analyzed (Participants) | 112 | 121
10^9/Litre
  Leukocytes, Baseline, n = 112, 121 | 6.8 (1.96) | 6.6 (1.97)
  Leukocytes, Week 36, n = 75, 98: number analyzed (Participants) | 75 | 98
  Leukocytes, Week 36, n = 75, 98 | 6.5 (1.81) | 6.5 (1.90)
  Platelets counts, Baseline, n = 112, 121 | 194.8 (48.79) | 204.4 (58.46)
  Platelets counts, Week 36, n = 75, 98: number analyzed (Participants) | 75 | 98
  Platelets counts, Week 36, n = 75, 98 | 193.3 (55.11) | 210.6 (73.28)

12. Secondary Outcome: Mean Values of Creatinine, Potassium, Phosphate, Parathyroid Hormone , Iron and Total Iron Binding Capacity Parameters at Baseline and Week 36
Description: Mean values of laboratory parameters: creatinine, potassium, phosphate, parathyroid hormone (PTH), iron and total iron binding capacity (TIBC) for each participant were estimated throughout the study. Summary data of mean values of laboratory parameters are presented at Baseline and Week 36.
Time Frame: Baseline and Week 36
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: micromoles per liter
Arm/Group | C.E.R.A. | Epoetin Alpha
Number analyzed (Participants) | 112 | 121
micromoles per liter
  Creatinine, Baseline, n = 109, 116: number analyzed (Participants) | 109 | 116
  Creatinine, Baseline, n = 109, 116 | 850.4 (242.22) | 916.6 (636.75)
  Creatinine, Week 36, n = 72, 95: number analyzed (Participants) | 72 | 95
  Creatinine, Week 36, n = 72, 95 | 881.0 (281.60) | 876.1 (265.33)
  Potassium, Baseline, n = 112, 121 | 5.2 (0.90) | 5.2 (0.83)
  Potassium, Week 36, n = 75, 99: number analyzed (Participants) | 75 | 99
  Potassium, Week 36, n = 75, 99 | 5.0 (0.74) | 5.0 (0.82)
  TIBC, Baseline, n = 60, 59: number analyzed (Participants) | 60 | 59
  TIBC, Baseline, n = 60, 59 | 37.0 (14.6) | 38.6 (10.23)
  TIBC, Week 36, n = 31, 43: number analyzed (Participants) | 31 | 43
  TIBC, Week 36, n = 31, 43 | 39.5 (15.4) | 39.4 (11.28)
  Iron, Baseline, n = 112, 121 | 14.2 (5.98) | 14.5 (6.12)
  Iron, Week 36, n = 73, 97: number analyzed (Participants) | 73 | 97
  Iron, Week 36, n = 73, 97 | 17.5 (7.94) | 12.5 (5.73)
  PTH, Baseline, n = 111, 121: number analyzed (Participants) | 111 | 121
  PTH, Baseline, n = 111, 121 | 228.3 (145.33) | 217.9 (158.57)
  PTH, Week 36, n = 18, 24: number analyzed (Participants) | 18 | 24
  PTH, Week 36, n = 18, 24 | 313.4 (297.39) | 368.2 (279.66)

13. Secondary Outcome: Mean Values of Albumin and Transferrin Concentration at Baseline and Week 36
Description: The mean values of albumin and transferrin concentration for each participant throughout the study was estimated. Summary data of mean values of albumin and transferrin concentration at baseline and week 36 are presented.
Time Frame: Baseline and Week 36
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: gram/litre
Arm/Group | C.E.R.A. | Epoetin Alpha
Number analyzed (Participants) | 111 | 118
gram/litre
  Albumin, Baseline, n = 111, 118 | 39.2 (4.14) | 39.9 (4.71)
  Albumin, Week 36, n = 72, 92: number analyzed (Participants) | 72 | 92
  Albumin, Week 36, n = 72, 92 | 39.3 (3.89) | 39.8 (4.57)
  Transferrin, Baseline, n = 56, 66: number analyzed (Participants) | 56 | 66
  Transferrin, Baseline, n = 56, 66 | 1.65 (0.38) | 1.77 (0.36)
  Transferrin, Week 36, n = 39, 49: number analyzed (Participants) | 39 | 49
  Transferrin, Week 36, n = 39, 49 | 1.76 (0.39) | 1.67 (0.33)

14. Secondary Outcome: Mean Values of Ferritin Concentration at Baseline and Week 36
Description: Mean values of ferritin concentration for each participant throughout the study was estimated. Summary data of mean values of ferritin concentration at Baseline and Week 36 are presented.
Time Frame: Baseline and Week 36
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: micrograms per liter
Arm/Group | C.E.R.A. | Epoetin Alpha
Number analyzed (Participants) | 112 | 121
micrograms per liter
  Ferritin, Baseline, n = 112,121 | 777.8 (529.23) | 621.4 (415.90)
  Ferritin, Week 36, n = 72, 93: number analyzed (Participants) | 72 | 93
  Ferritin, Week 36, n = 72, 93 | 736.9 (467.00) | 609.9 (379.53)

15. Secondary Outcome: Mean Values of Transferrin Saturation at Baseline and Week 36
Description: The mean values of transferrin saturation (TS) for each participant were estimated throughout the study. Summary data of mean values of TS at Baseline and Week 36 are presented.
Time Frame: Baseline and Week 36
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | C.E.R.A. | Epoetin Alpha
Number analyzed (Participants) | 112 | 121
percentage
  TS, Baseline; n = 112, 121 | 38.0 (17.32) | 36.2 (17.96)
  TS, Week 36; n = 70, 91: number analyzed (Participants) | 70 | 91
  TS, Week 36; n = 70, 91 | 44.4 (23.64) | 31.7 (18.72)

16. Secondary Outcome: Mean Values of Aspartate Transaminase and Alkaline Phosphatase at Baseline and Week 36
Description: The mean values of aspartate transaminase (AST) and alkaline phosphatase (ALP) levels in serum for each participant were estimated throughout the study. Summary data of mean values of Potassium and alkaline phosphatase level in serum at Baseline and Week 36 are presented.
Time Frame: Baseline and Week 36
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: International units/Liter
Arm/Group | C.E.R.A. | Epoetin Alpha
Number analyzed (Participants) | 109 | 119
International units/Liter
  AST, Baseline, n = 109, 117: number analyzed (Participants) | 109 | 117
  AST, Baseline, n = 109, 117 | 16.4 (7.48) | 16.6 (8.09)
  AST, Week 36, n = 74, 96: number analyzed (Participants) | 74 | 96
  AST, Week 36, n = 74, 96 | 17.2 (10.07) | 17.1 (12.47)
  ALP, Baseline, n = 108, 119: number analyzed (Participants) | 108 | 119
  ALP, Baseline, n = 108, 119 | 106.4 (51.01) | 118.0 (73.44)
  ALP, Week 36, n = 73, 93: number analyzed (Participants) | 73 | 93
  ALP, Week 36, n = 73, 93 | 116.2 (77.4) | 129.7 (84.99)

17. Secondary Outcome: Number of Participants With Adverse Events and Serious Adverse Events
Description: An adverse event (AE) was defined as any untoward medical occurrence in a subject who is administered a study treatment regardless of whether or not the event has a causal relationship with the treatment. An AE, therefore, could be any unfavorable or unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the study treatment, whether or not related to the treatment. A Serious Adverse Event (SAE) is any untoward medical occurrence that at any dose results in death, are life threatening, requires hospitalization or prolongation of hospitalization or results in disability/incapacity, and congenital anomaly/birth defect. Number of participants with at least one AE and SAE were reported.
Time Frame: Up to Week 40
Population: The analysis was performed on Safety Population.
Measure: Number; unit: participants
Arm/Group | C.E.R.A. | Epoetin Alpha
Number analyzed (Participants) | 112 | 121
participants
  Any AE | 99 | 106
  Any SAE | 27 | 16

18. Secondary Outcome: Number of Participants With Abnormal Changes in ECG From Baseline to Week 40
Description: Twelve-lead ECG was performed.
Time Frame: From Baseline to Week 40
Population: The analysis was performed on Safety population.
Measure: Number; unit: participants
Arm/Group | C.E.R.A. | Epoetin Alpha
Number analyzed (Participants) | 112 | 121
participants | 0 | 0

19. Secondary Outcome: Number of Participants With Abnormal Changes in Vital Signs From Baseline to Week 40
Description: Vital signs included blood pressure, pulse rate and body weight.
Time Frame: From Baseline to Week 40
Population: The analysis was performed on safety population.
Measure: Number; unit: participants
Arm/Group | C.E.R.A. | Epoetin Alpha
Number analyzed (Participants) | 112 | 121
participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to Week 40 (follow up)
Description: The adverse events were reported in safety analysis population. The safety analysis population included those participants who have been treated with at least one dose of the trial medication and a safety follow-up, whether withdrawn prematurely or not.
Arm/Group | C.E.R.A. | Epoetin Alpha
Serious Adverse Events (participants affected / at risk) | 27/112 | 16/121
Other Adverse Events (participants affected / at risk) | 83/112 | 92/121
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | C.E.R.A. (N=112) | Epoetin Alpha (N=121)
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Coagulopathy (Blood and lymphatic system disorders) | 0 | 1
Acute Myocardial Infarction (Cardiac disorders) | 1 | 0
Angina Unstable (Cardiac disorders) | 1 | 0
Atrial Fibrillation (Cardiac disorders) | 1 | 0
Myocardial Infarction (Cardiac disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Duodenal ulcer (Gastrointestinal disorders) | 1 | 0
Gastric Haemorrhage (Gastrointestinal disorders) | 0 | 1
Upper Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 2 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Chest pain (General disorders) | 2 | 0
Sudden death (General disorders) | 0 | 1
Cholestasis (Hepatobiliary disorders) | 1 | 0
Hepatic failure (Hepatobiliary disorders) | 1 | 0
Hypersensitivity (Immune system disorders) | 0 | 1
Appendicitis (Infections and infestations) | 1 | 0
Endocarditis (Infections and infestations) | 1 | 0
Infection (Infections and infestations) | 0 | 1
Lung Infection (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 4 | 4
Postoperative Wound Infection (Infections and infestations) | 1 | 0
Respiratory Tract Infection (Infections and infestations) | 0 | 1
Urinary Tract Infection (Infections and infestations) | 1 | 0
Arteriovenous Fistula Aneurysm (Injury, poisoning and procedural complications) | 0 | 1
Arteriovenous Fistula Thrombosis (Injury, poisoning and procedural complications) | 2 | 0
Lower Limb Fracture (Injury, poisoning and procedural complications) | 1 | 0
Renal Haematoma (Injury, poisoning and procedural complications) | 0 | 1
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 1
Haemoglobin Decreased (Investigations) | 1 | 0
Diabetic foot (Metabolism and nutrition disorders) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0
Hypervolaemia (Metabolism and nutrition disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Convulsion (Nervous system disorders) | 1 | 1
Haemorrhagic Stroke (Nervous system disorders) | 0 | 1
Ischaemic Stroke (Nervous system disorders) | 0 | 1
Metrorrhagia (Reproductive system and breast disorders) | 1 | 0
Acute Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonia Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Skin Ulcer (Skin and subcutaneous tissue disorders) | 1 | 0
Aortic Dissection (Vascular disorders) | 0 | 1
Deep Vein Thrombosis (Vascular disorders) | 1 | 1
Hypertensive Crisis (Vascular disorders) | 2 | 0
Hypotension (Vascular disorders) | 1 | 0
Varicose vein (Vascular disorders) | 1 | 0
Localised Infection (Infections and infestations) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | C.E.R.A. (N=112) | Epoetin Alpha (N=121)
Abdominal pain (Gastrointestinal disorders) | 11 | 13
Abdominal pain upper (Gastrointestinal disorders) | 5 | 9
Diarrhoea (Gastrointestinal disorders) | 14 | 9
Dyspepsia (Gastrointestinal disorders) | 1 | 7
Gastritis (Gastrointestinal disorders) | 6 | 5
Nausea (Gastrointestinal disorders) | 8 | 6
Vomiting (Gastrointestinal disorders) | 8 | 2
Chest pain (General disorders) | 8 | 7
Malaise (General disorders) | 9 | 4
Influenza (Infections and infestations) | 1 | 10
Respiratory Tract Infection (Infections and infestations) | 6 | 5
Upper Respiratory Tract Infection (Infections and infestations) | 5 | 8
Urinary Tract Infection (Infections and infestations) | 5 | 7
Arteriovenous Fistula Site Complication (Injury, poisoning and procedural complications) | 6 | 5
Arteriovenous Fistula Thrombosis (Injury, poisoning and procedural complications) | 6 | 5
Hyperphosphataemia (Metabolism and nutrition disorders) | 3 | 7
Hypervolaemia (Metabolism and nutrition disorders) | 7 | 2
Hypoglycaemia (Metabolism and nutrition disorders) | 5 | 7
Back Pain (Musculoskeletal and connective tissue disorders) | 9 | 16
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 23 | 17
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 8 | 11
Dizziness (Nervous system disorders) | 6 | 6
Headache (Nervous system disorders) | 12 | 24
Cough (Respiratory, thoracic and mediastinal disorders) | 9 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 8 | 6
Hypertension (Vascular disorders) | 18 | 15
Hypotension (Vascular disorders) | 19 | 20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.